CLINICAL TRIAL: NCT01240642
Title: A Multi-center, Open-label, Dose-escalation Study in Patients With Advanced Cacner to Determine the Effect of the ASA404 Infusion Rate and Co-administration With the Paclitaxel Plus Carboplatin Regimen or Docetaxel on the Pharmacokinetics of Free and Total ASA404
Brief Title: An Open-label, Dose Escalation Multi-center Study in Patients With Advanced Cancer to Determine the Infusion Rate Effect of ASA 404 With Paclitaxel Plus Carboplatin Regimen or Docetaxel on the Pharmacokietics of Free and Total ASA404
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASA404A2112; EudraCT 2009-011142-26 (Registry Identifier: EudraCT)
Record Dates: First submitted 2010-11-11; First posted 2010-11-15 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2012-11

CONDITIONS: Metastatic Cancer With Impaired Renal Function; Metastatic Cancer With Normal Renal Function
Keywords: Advanced or metastatic cancer; refractory; core phase; extension phase; dose escalation; standard chemotherapy; doctaxel; paclitaxel; carboplatin; safety; tolerability
MeSH Terms: conditions — Neoplasm Metastasis | interventions — vadimezan

ARMS (1):
- ASA404 (Experimental)
  Interventions: Drug: ASA404

INTERVENTIONS:
Drug: ASA404

SUMMARY:
The purpose of this study is to determine the effect of the ASA404 infusion rate and co-administrating ASA404 with paclitaxel + carbopaltin chemotherapy regimen or docetaxel on the pharamcokinetics (PK) of free and total ASA404.

ELIGIBILITY:
Inclusion Criteria:

* Patients having histologically-proven solid tumors, who are either refractory to standard chemotherapy
* Patients whom chemotherapy with an investigaional agent in combination with docetaxel, or paclitaxel + carboplatin is appropriate
* Creatinine clearance according to Cockcroft-Gault formula : Normal > 80 mL/min, Mild 50-80 mL/min, Moderate 30-<50 mL/min
* A minimum of 4 weeks must have elapsed since the last treatment with other cancer therapies
* Potassium, calcium, magnesium and phosphorus values within the normal range
* Body Mass Index (BMI) must be within the range of 18 and 30

Exclusion Criteria:

* Patients having CNS metastases, must have a CT or MRI of the brain performed to rule out CNS metastases
* Patients with leptomeningeal disease metastases
* Radiotherapy </- weeks prior to starting study drug
* Major surgery </ 4 weeks prior to the start of study
* Administration of CYP1A2 and CYP3A4/5 enzyme inducing or inhibiting drugs within 14 days prior to starting study drug

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the pK of a single intravenous dose of ASA404 1200 and 1800 mg/m2 monotherapy in adult cancer patients with impaired renal function compared to matching patients with normal renal function | 12 monnths

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of a single i.v. dose of ASA 1200 and 1800 mg/m2 +chemotherapy (doctaxel or paclitaxel + carboplatin) in adult cancer patients with impaired renal function compared to matching patients with normal renal function | 12 months
To assess the safety and tolerability of ASA404 in adult cancer patients with impaired renal function compared to matching patients with normal renal function | 12 months
To assess the safety and tolerability of ASA404 1200 or 1800 mg/m2 in combination with chemotherapy (docetaxel or paclitaxel + carboplatin) | 12 months
To evaluate ASA404 pharmacokinetic parameters including AUC (0-t last),), AUC (0-inf)), T ((½)), CL, V(Z), Cmax, and Tmax | 12 months
To evaluate renal clearance (CLR) of ASA404. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Belgium (4):
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Jette
  - Novartis Investigative Site, Saint-Lambert
  - Novartis Investigative Site, Wilrijk

REFERENCES:
- See also: Results for CASA404A2112 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=5424